CLINICAL TRIAL: NCT02702557
Title: Feasibility Study of Unsupervised Elastic Band Exercises Performed by Frail Elderly Hospitalized Patients Monitored by the Bandcizer as a Supplement to Usual Supervised Physiotherapy Sessions
Brief Title: Unsupervised Elastic Band Exercises Performed by Frail Elderly Hospitalized Patients Monitored by the Bandcizer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Collaborators: Aalborg University (Other); Amager Hospital (Other); Hvidovre University Hospital (Other); University of Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2016-42
Record Dates: First submitted 2016-02-29; First posted 2016-03-08 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-05

CONDITIONS: Frail Elderly
Keywords: Frail Elderly; Elastic Band Exercises; Unsupervised Exercises; Monitoring Technology; Bandcizer; Adherence; Feasibility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Elastic Band Exercises (Other): Unsupervised Elastic band exercises performed once a day until the patient is discharged from the hospital. One exercise for the upper extremity (row exercise level 1-3) and one exercise for the lower extremity (knee extension level 1-3). The two exercises are both performed as 3 sets of 10 repetitions.
  Interventions: Other: Elastic Band Exercises

INTERVENTIONS:
Other: Elastic Band Exercises
  Other Names: Bandcizer

SUMMARY:
This feasibility study investigates if frail elderly and hospitalized patients are able to perform unsupervised elastic band exercises as a supplement to their usual supervised physiotherapy sessions and how much training they perform during their hospitalization. It is also investigated how the frail elderly and the health personnel experiences the unsupervised elastic band exercises.

ELIGIBILITY:
Inclusion Criteria:

* Frail elderly and hospitalized patients with a minimal score of 5/15 measured by the Tilburg Frailty Indicator
* Able to read and understand Danish

Exclusion Criteria:

* Frail elderly and hospitalized patients with a score of <5 measured by the Short Portable Mental Status Questionnaire
* Frail elderly and hospitalized patients where resistance training and physical activity is contraindicated (evaluated by a geriatrician and/or physiotherapist)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-02; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Total number of sets performed | From inclusion-discharge from hospital - up to 6 weeks

SECONDARY OUTCOMES:
The total number of repetitions performed | From inclusion-discharge from hospital - up to 6 weeks

OTHER OUTCOMES:
Mean deviation from the prescribed TUT per repetition in seconds during the course of the intervention | From inclusion-discharge from hospital - up to 6 weeks
  The mean deviation is calculated as the difference between actual TUT and prescribed TUT (8 seconds).
Difference in score of two tests: The 30-s chair stand and the de Morton Mobility Index (DEMMI) | From beginning of hospitalization to discharge from hospital - up to 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jane Andreasen, ph.d. stud., Principal Investigator — Department of Occupational Therapy and Physiotherapy, Aalborg University Hospital
Locations (1):
- Aalborg University Hospital, Aalborg, North Region Denmark, Denmark

REFERENCES:
- [Derived] Rathleff CR, Bandholm T, Spaich EG, Jorgensen M, Andreasen J. Unsupervised progressive elastic band exercises for frail geriatric inpatients objectively monitored by new exercise-integrated technology-a feasibility trial with an embedded qualitative study. Pilot Feasibility Stud. 2017 Nov 13;3:56. doi: 10.1186/s40814-017-0202-3. eCollection 2017. PMID 29158914